CLINICAL TRIAL: NCT02754661
Title: Multicenter, Prospective, Randomized Study Comparing the Diagnostic Yield of Colon Capsule Endoscopy Versus Computed Tomographic Colonography in a Screening Population
Brief Title: Colon Capsule Endoscopy (CCE) Versus Computed Tomographic Colonography (CTC) in the Identification of Colonic Polyps in a Screening Population.
Acronym: TOPAZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COVGIC20543; MA-213 (Other: Medtronic)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer Screening
Keywords: Polyps; Capsule endoscopy; CT Colonography; Colonoscopy; Average risk patients for colorectal cancer screening
MeSH Terms: conditions — Polyps | interventions — Endoscopy; Colonography, Computed Tomographic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- COLON Capsule endoscopy (Experimental): Subjects will be instructed to follow a detailed dietary and colon preparation regimen prior to and during the CCE procedure day. With the exception of Gastrografin, all colon preparation products will be standard colon cleansing products approved by the FDA.
  Between 45 and 75 minutes after the final Polyethylene Glycol (PEG) ingestion, the subject will swallow the PillCam COLON Capsule with a cup of water.
  If necessary, capsule position will be monitored to ensure adequate booster administration. Subjects will keep a timed diary of key preparation steps and bowel activity, including capsule excretion. Subjects will be allowed to leave the unit 10 hours after capsule ingestion if the capsule is not yet excreted. Subjects leaving before excretion will be instructed to disconnect the recorder at excretion or 12 hours after capsule ingestion (whichever comes first).
  Interventions: Device: COLON Capsule endoscopy
- Computed Tomographic Colonography (Active Comparator): Subjects will be instructed to follow a detailed dietary and colon preparation regimen prior to and during the Computed Tomographic Colonography (CTC) procedure day.
  The CTC procedure and study interpretation will be conducted in accordance with the ACR-SAR-SCBT-MR Practice Parameter for the Performance of CT Colonography in Adults. Colon insufflation will be performed with the subject in the lateral decubitus or supine position.With the subject in the supine position, a CT scout image will be taken to confirm adequate colon distention. If adequate bowel distention is not achieved, additional air will be insufflated into the colon. After scanning the subject in the supine position, the subject will be placed in the prone position, and additional CO2 will be administered. Subsequently, CT will be performed with the subject in the prone position. If a prone position is not possible for the subject, a left lateral decubitus position is preferred for optimal gas and fluid redistribution.
  Interventions: Device: Computed Tomographic Colonography

INTERVENTIONS:
Device: COLON Capsule endoscopy
  Arms: COLON Capsule endoscopy
Device: Computed Tomographic Colonography
  Arms: Computed Tomographic Colonography

SUMMARY:
The primary objective of this multicenter, prospective, randomized study is to assess the diagnostic yield of Colon Capsule Endoscopy (CCE) versus Computed Tomographic Colonography (CTC) in a screening population.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized study to evaluate the efficacy of CCE versus CTC in the identification of colonic polyps in a screening population.

Subjects will be enrolled at up to 20 clinical sites in the United States. Subjects who meet the eligibility criteria will be screened by the gastroenterology site for study participation at a baseline visit which will also include a blood test for renal function (eGFR), and will be evaluated on the randomized procedure day (CCE versus CTC) and again on the day of both the blinded and unblinded OC procedures. Telephone follow-ups will be conducted 5 - 9 days after the CCE/CTC procedure and 5 - 9 days after the unblinded OC procedure to assess subject well-being and capture any Adverse Events (AEs), regardless of relationship to the CCE, CTC, or Optical colonoscopy (OC) procedures.

All CCE RAPID® videos and CTC images will be evaluated by local and central readers. All study analyses will be based on central reader results for both CCE and CTC. Two sets of central readers will be utilized, one set for reading of the CCE RAPID® videos and one set for reading the CTC studies. Both groups of readers will be experts in the reading process for their respective procedures. Readers will provide a report of their findings to the sponsor within 2 weeks of capsule ingestion or CTC procedure in order to allow subjects to return within 5 weeks capsule ingestion or CTC procedure to undergo confirmatory OC. The first OC procedure will be performed with the clinician blinded to the CCE or CTC results. Immediately following this blinded procedure, the clinician will review the CCE or CTC results report provided by the sponsor from the central readers, and a second unblinded OC procedure will be performed if there are discrepancies between the CCE/CTC findings and OC.

Colonoscopy must not be performed by the same person who conducts the local CCE reading, or anyone who has reviewed CCE/CTC results for that subject.

Bowel preparation regimens for all three procedure types will be standardized across sites.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 and 75 years of age (for African Americans only, subject is between 45-75 years of age).
2. Subject is classified as average risk per the American Gastroenterological Association Guidelines on Colorectal Cancer Screening: Individuals without a personal or family history of CRC or adenomas, inflammatory bowel disease, or high-risk genetic syndromes.
3. Subject is willing and able to participate in the study procedures and to understand and sign the informed consent.

Exclusion Criteria:

1. Subject with history of colorectal cancer or adenoma (including those identified by computed tomography [CT], optical colonoscopy [OC[, sigmoidoscopy, etc.).
2. Subject with history of negative colonoscopy within 10 years, as these subjects would be defined as not requiring screening in this timeframe. For subjects with alternative screening methods, refer to applicable guidelines.
3. Subject with currently suspected or diagnosed with hematochezia, melena, iron deficiency with or without anemia, or any other rectal bleeding, including positive fecal occult blood test of any variety.
4. Subject with any current condition believed to have an increased risk of capsule retention such as suspected or known bowel obstruction, stricture, or fistula.
5. Subject with current dysphagia or any swallowing disorder.
6. Subject with current serious medical conditions that would increase the risk associated with CCE, CTC, or colonoscopy that are so severe that screening would have no benefit.
7. Subject with a cardiac pacemaker or other implanted electromedical device.
8. Subject expected to undergo MRI examination within 7 days after ingestion of the capsule.
9. Subject with clinical evidence of renal disease, including clinically significant laboratory abnormalities of renal function within the past 6 months, or at any time in the past if not tested within the last 6 months, defined as creatinine, blood urea nitrogen (BUN), and/or glomerular filtration rate (GFR) outside of the local laboratory reference range.
10. Subject with a diagnosis of gastroparesis or small bowel or large bowel dysmotility.
11. Subject with allergies or known contraindication to the medications or preparation agents used in the procedure as described in the relevant instructions for use.
12. Subject has an estimated life expectancy of less than 6 months.
13. Subject is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).
14. Subject is pregnant, suspected pregnant, or is actively breast-feeding. Females of child-bearing potential will be required to provide either a urine pregnancy test or serum pregnancy test as part of the participant's standard of care regardless of their participation in the study (except for subjects who are surgically sterile or are post-menopausal for at least two years).
15. Subject has participated in an investigational drug or device research study within 30 days of enrollment that may interfere with the subject's safety or ability to participate in this study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Cash, MD, Principal Investigator — University of South Alabama
Locations (13):
- United States (13):
  - University of South Alabama, Mobile, Alabama
  - Borland-Groover Clinic, Jacksonville, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Indianapolis Gastroenterology and Hepatology, Indianapolis, Indiana
  - Baystate Hospital, Springfield, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Clinical Research Professionals, St Louis, Missouri
  - NYU, New York, New York
  - Columbia University, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Virginia Gastroenterology institute, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cash BD, Fleisher MR, Fern S, Rajan E, Haithcock R, Kastenberg DM, Pound D, Papageorgiou NP, Fernandez-Urien I, Schmelkin IJ, Rex DK. Multicentre, prospective, randomised study comparing the diagnostic yield of colon capsule endoscopy versus CT colonography in a screening population (the TOPAZ study). Gut. 2021 Nov;70(11):2115-2122. doi: 10.1136/gutjnl-2020-322578. Epub 2020 Dec 18. PMID 33443017

RESULTS

PARTICIPANT FLOW:
Groups:
- COLON Capsule Endoscopy: Subjects who had Colon capsule followed by optical colonoscopy within 5-6 weeks.
- Computed Tomographic Colonography: Subjects who had computed Tomographic Colonography followed by optical colonoscopy within 5-6 weeks.
Period: Overall Study
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
Started | 160 | 160
Completed | 145 | 141
Not Completed | 15 | 19

BASELINE CHARACTERISTICS:
Population: Baseline Analysis population is based on the Full Analysis set defined as all randomized subjects who underwent colonoscopy and CTC or CCE procedures.
Groups:
- COLON Capsule Endoscopy: Subjects who had colon capsule endoscopy followed by optical colonoscopy within 5-6 weeks.
- Total: Total of all reporting groups
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography | Total
Number analyzed (Participants) | 145 | 141 | 286
Age, Customized [Mean (Full Range); unit: year] | 55.3 [46.1 to 73.9] | 56.0 [45.8 to 75.5] | 55.7 [45.8 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 73 | 165
  Male | 53 | 68 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 138 | 133 | 271
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 23 | 56
  White | 109 | 115 | 224
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 145 | 141 | 286
BMI (Body Mass Index) [Mean (Full Range); unit: kg/m^2] | 32.2 [18.5 to 67.9] | 30.2 [18.2 to 52.5] | 31.2 [18.2 to 67.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Actionable Lesion on CCE vs. CTC Confirmed by Optical Colonoscopy
Description: Proportion of subjects shown to have an actionable lesion, defined as any polyp or mass lesion ≥6 mm.
  Diagnostic yield of CCE/CTC will be calculated in relation to the confirmatory Optical colonoscopy results
Time Frame: 5-6 weeks from randomized procedure
Population: Per protocol Analysis set (PPAS) is comprised of randomized subjects without major protocol deviations (violations with significant impact on subject outcomes) and who don't meet any of the following criteria: Subject withdraws, Capsules remained in the stomach/SB during the entire procedure, colonoscopy could not be done, technical failure
Measure: Count of Participants; unit: Participants
Arm/Group | COLON CAPSULE ENDOSCOPY | Computed Tomographic Colonography
Number analyzed (Participants) | 133 | 128
Participants | 34 | 11
Statistical Analysis 1: Comparison: COLON CAPSULE ENDOSCOPY vs Computed Tomographic Colonography; Test type: Non-Inferiority — The non-inferiority margin (δ) is pre-defined to be 5% in this study. Posterior Probability was based on Bayesian analysis; Posterior Probability Bayesian analysis = 0.9999 — Support the claim of statistical non-inferiority of CCE vs CTC

2. Secondary Outcome: Sensitivity of CCE Versus CTC in the Detection of Polyps ≥6 mm
Description: Sensitivity (the percentage of patients with disease who test positive) assessed in relation to the confirmatory optical colonoscopy (OC) results on a "per subject" basis
Time Frame: 5-6 weeks from randomized procedure
Population: Per protocol Analysis (PPAS) set is comprised of randomized subjects without major protocol deviations (violations with significant impact on subject outcomes) and who don't meet any of the following criteria: Subject withdraws, Capsules remained in the stomach/SB during the entire procedure, colonoscopy could not be done, technical failure
Measure: Count of Participants; unit: Participants
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
Number analyzed (Participants) | 53 | 41
Participants | 34 | 11
Statistical Analysis 1: Comparison: COLON Capsule Endoscopy vs Computed Tomographic Colonography; Test type: Non-Inferiority — Non-inferiority margin was set as 10%; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 0.3732, 90% CI 2-sided [0.2030 to 0.5434] — Based on Farrington-Manning Method

3. Secondary Outcome: Specificity of CCE Versus CTC in the Detection of Polyps ≥6 mm
Description: Specificity (the percentage of patients without disease who test negative) assessed in relation to the confirmatory optical colonoscopy (OC) results on a "per subject" basis
Time Frame: 5-6 weeks from randomized procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
Number analyzed (Participants) | 80 | 87
Participants | 77 | 86
Statistical Analysis 1: Comparison: COLON Capsule Endoscopy vs Computed Tomographic Colonography; Test type: Non-Inferiority — Non-inferiority margin was set as 10%; p = 0.0190, Farrington-Manning test; Risk Difference (RD) = -0.026, 90% CI 2-sided [-0.0847 to 0.0327] — Based on Farrington-Manning Method

4. Secondary Outcome: Predictive Value of a Positive Test (PPV) of CCE Versus CTC in the Detection of Polyps ≥6 mm
Description: Predictive value of a positive test (PPV) is the percentage of patients with positive tests who have disease assessed in relation to the confirmatory OC results on a "per subject" basis
Time Frame: 5-6 weeks from randomized procedure
Population: Per protocol Analysis set is comprised of all randomized subjects without major protocol deviations (violations that may have a significant impact on subject outcomes) and who don't meet any of the following criteria: Subject withdraws, Capsules remained in the stomach/SB during the entire procedure, colonoscopy could not be done, technical failure
Measure: Count of Participants; unit: Participants
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
Number analyzed (Participants) | 37 | 12
Participants | 34 | 11
Statistical Analysis 1: Comparison: COLON Capsule Endoscopy vs Computed Tomographic Colonography; Test type: Non-Inferiority — Non-inferiority margin was set as 10%; p = 0.0930, Farrington-Manning test; Risk Difference (RD) = 0.0023, 90% CI 2-sided [-0.1249 to 0.1249] — Based on Farrington-Manning Method

5. Secondary Outcome: Predictive Value of a Negative (NPV) of CCE Versus CTC in the Detection of Polyps ≥6 mm
Description: Predictive value of a negative test (NPV) is the percentage of patients with negative tests who do not have disease, assessed in relation to the confirmatory OC results on a "per subject" basis.
Time Frame: 5-6 weeks from randomized procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
Number analyzed (Participants) | 96 | 116
Participants | 77 | 86
Statistical Analysis 1: Comparison: COLON Capsule Endoscopy vs Computed Tomographic Colonography; Test type: Non-Inferiority — Non-inferiority margin was set as 10%; p = 0.0034, Farrington-Manning test; Risk Difference (RD) = 0.0607, 90% CI 2-sided [-0.0371 to 0.1585] — Based on Farrington-Manning Method

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 5-6 week period
Description: Adverse events have been collected at the start of the CCE/CTC bowel preparation up until colonoscopy Follow-up call. The following AEs and serious adverse events (SAEs) were collected:
  * All adverse events related to the CCE, CTC and or OC procedures
  * All retained capsules greater than 14 days
  * All perforations
  * All device deficiencies that may lead to a SAE
  * All adverse events that meet serious adverse event definition
  * All deaths
Arm/Group | COLON Capsule Endoscopy | Computed Tomographic Colonography
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/141
Serious Adverse Events (participants affected / at risk) | 2/145 | 1/141
Other Adverse Events (participants affected / at risk) | 4/145 | 8/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COLON Capsule Endoscopy (N=145) | Computed Tomographic Colonography (N=141)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0
Rectal Haemorrage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post procedural haemorrahage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COLON Capsule Endoscopy (N=145) | Computed Tomographic Colonography (N=141)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemmorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02754661/Prot_SAP_000.pdf